CLINICAL TRIAL: NCT05981846
Title: A Phase II, Randomized, Double-blind, Multi-centre Trial to Evaluate the Safety and Immunogenicity of BIMERVAX® When Coadministered With Seasonal Surface Antigen, Inactivated, Adjuvanted Influenza Vaccine (SIIV) in Adults Older Than 65 Years of Age Fully Vaccinated Against COVID-19
Brief Title: A Phase II Trial to Evaluate the Safety and Immunogenicity of BIMERVAX® When Coadministered With Seasonal Influenza Vaccine (SIIV) in Adults Older Than 65 Years of Age Fully Vaccinated Against COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hipra Scientific, S.L.U (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HIPRA-HH-11
Record Dates: First submitted 2023-08-07; First posted 2023-08-08 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: SARS CoV 2 Infection; Influenza, Human
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BIMERVAX + SIIV (Experimental)
  Interventions: Biological: BIMERVAX; Biological: SIIV
- BIMERVAX + PLACEBO (Active Comparator)
  Interventions: Biological: BIMERVAX
- SIIV + PLACEBO (Active Comparator)
  Interventions: Biological: SIIV

INTERVENTIONS:
Biological: BIMERVAX — One dose of booster vaccine
  Arms: BIMERVAX + PLACEBO; BIMERVAX + SIIV
Biological: SIIV — One dose
  Arms: BIMERVAX + SIIV; SIIV + PLACEBO

SUMMARY:
This is a Phase II, randomized, double-blind, multi-centre trial to evaluate the safety and immunogenicity of BIMERVAX® when coadministered with seasonal surface antigen inactivated adjuvanted influenza vaccine (SIIV) in adults older than 65 years of age fully vaccinated against COVID-19.

In this study approximately 300 adults aged 65 or older will be enrolled and followed for 1 month after study treatment. Safety and immunogenicity of all participants will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 65 or older at Day 0.
2. Are willing and able to sign the informed consent and can comply with all study visits and procedures.
3. Participant must have received at least a primary scheme of an mRNA vaccine (2 doses). Booster doses or previous COVID-19 infections are allowed. Last dose must have been administered at least 6 months before Day 0. History of COVID-19 infection is allowed if occurred at least >30 days before Day 0.
4. Have a negative Rapid Antigen Test (RAT) at Day 0 before vaccinations.
5. Adults determined by clinical assessment, including medical history and clinical judgement, to be eligible for the study, including adults with pre-existing chronic and stable diseases (non-immunocompromised), if these are stable and well-controlled according to the investigator's judgment.

   Exclusion Criteria:
6. Acute illness with fever ≥ 38.0°C at Day 0 or within 24 hours prior to vaccination. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator.
7. Allergy to egg proteins (egg or egg products) or chicken proteins.
8. History of Guillain-Barré syndrome (GBS)
9. History of COVID-19 infection (described as a positive RAT or PCR), in the previous 30 days before Day 0.
10. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behaviour that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
11. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g. anaphylaxis) to any component of the study intervention(s).
12. Immunocompromised individuals defined as those with primary and secondary immune deficiencies and those receiving chemotherapy or immunosuppressant drugs other than steroids and glucocorticoids (maximum 30mg/day of prednisone, or equivalent, by any administration route for a maximum of 30 consecutive days), within 90 days prior to vaccination or during the study.
13. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
14. Receipt of blood-derived immune globulins, blood, or blood-derived products in the past 3 months.
15. Participation in other studies involving study intervention within 28 days prior to screening and/or during study participation.
16. Received any non-study vaccine within 14 days before or after screening. For live or attenuated vaccines, 4 weeks before or after screening.
17. History of a diagnosis or other conditions that, in the judgment of the investigator, may affect study endpoint assessment or compromise participant safety.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 279 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Number, percentage, and characteristics of solicited local and systemic reactions through Day 7 after vaccination. | Day 0, Day 7
Number, percentage, and characteristics of unsolicited local and systemic adverse events (AEs) through the end of the study. | Day 0, Day 7, Day 28
Number and percentage of serious adverse events (SAEs) through the end of the study. | Day 0, Day 7, Day 28
Number and percentage of adverse events of special interest (AESI) through the end of the study | Day 0, Day 7, Day 28

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - CAP Centelles, Centelles, Barcelona
  - Hospital HM Modelo, A Coruña
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Josep Trueta, Girona
  - Hospital Regional de Málaga, Málaga
  - Hospital Clínico de Valladolid, Valladolid